CLINICAL TRIAL: NCT07232550
Title: Biomarkers and Respiratory Omics as New CHildren Opportunities - Study of Clinical Outcomes and Predictivity Evaluation - a Multi-cohort, Multi-center Study
Brief Title: Biomarkers and Respiratory Omics as New CHildren Opportunities - Study of Clinical Outcomes and Predictivity Evaluation
Acronym: BRONCHOSCOPE
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: Medical University of Lodz (Other); Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: KB/100/2025
Record Dates: First submitted 2025-09-25; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Asthma in Children; Protracted Bacterial Bronchitis; Chronic Cough
Keywords: PBB; Asthma
MeSH Terms: conditions — Chronic Cough; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage fluid; sputum; mucosal biopsy; whole blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Asthma: Children diagnosed with asthma at the baseline
  Interventions: Procedure: fiberoptic bronchoscopy; Procedure: blood sample collection; Diagnostic Test: Respiratory functional tests; Diagnostic Test: Sputum culture
- Protracted Bacterial Bronchitis: Children diagnosed with Protracted Bacterial Bronchitis at the baseline
  Interventions: Procedure: fiberoptic bronchoscopy; Procedure: blood sample collection; Diagnostic Test: Respiratory functional tests; Diagnostic Test: Sputum culture
- Children without asthma who have been exposed to inhaled glucocorticosteroids: Children without asthma who have been exposed to inhaled glucocorticosteroids for at least 4 weeks during the 2 months preceeding bronchoscopy
  Interventions: Procedure: fiberoptic bronchoscopy; Procedure: blood sample collection; Diagnostic Test: Respiratory functional tests; Diagnostic Test: Sputum culture
- Non inflammatory causes of chronic cough: Children diagnosed with: laryngomalacia, tracheobronchomalacia adenoid hypertrophy, gastroesophageal reflux disease, habitual cough
  Interventions: Procedure: fiberoptic bronchoscopy; Procedure: blood sample collection; Diagnostic Test: Respiratory functional tests; Diagnostic Test: Sputum culture
- Control group: Children without underlying diseases who undergo bronchoscopy either for suspected foreign body aspiration or as part of routine diagnostic evaluation
  Interventions: Procedure: fiberoptic bronchoscopy; Procedure: blood sample collection; Diagnostic Test: Respiratory functional tests; Diagnostic Test: Sputum culture

INTERVENTIONS:
Procedure: fiberoptic bronchoscopy — During procedure performing physician will evaluate respiratory tract anatomy. Samples of bronchoalveolar lavage fluid will be collected for culture, cellular composition analysis, amphiregulin level, cytokine profiling, metagenomic sequencing, metabolomic assessment, additionally mucosal biopsy will be performed using forceps and brush techniques for histopathological evaluation
Procedure: blood sample collection — 5 mL sample of blood will be collected in each individual at baseline and during follow-up visits for complete blood count and Immunoglobulin E levels
Diagnostic Test: Respiratory functional tests — At baseline and during each follow-up visit children will perform spirometry, Impulse Oscillometry and Fractional Exhaled Nitric Oxide
Diagnostic Test: Sputum culture — At baseline and during first follow-up visit sputum will be collected from each individual for culture

SUMMARY:
The goal of this observational study is to improve the identification of biomarkers that predict disease progression and to assess the effectiveness of current therapies in children with asthma and protracted bacterial bronchitis.

The main aim of the study is to evaluate the microbiome composition and diversity, cellular composition, and metabolomic profile. In addition, to assess their correlation on subsequent treatment and disease course in children with asthma, protracted bacterial bronchitis, and in those receiving inhaled glucocorticosteroids without a diagnosis of asthma.

Participants will undergo fiberoptic bronchoscopy. During bronchoscopy, the performing physician will collect Bronchoalveolar lavage fluid samples for metagenomic and metabolomic analysis, as well as mucosal biopsies for histopathological evaluation.

DETAILED DESCRIPTION:
This prospective cohort study will enroll 160 participants and allocate them into study arms according to their medical history. The planned arms include: children with asthma, children with protracted bacterial bronchitis, children without asthma who are exposed to inhaled glucocorticosteroids, children with chronic cough, and a control group.

Participants will be recruited from the Pediatric Pulmonology Departments of the Medical Universities in Warsaw and Lodz. At baseline, investigators will administer a standardized medical questionnaire approved by both medical centers. All participants will undergo a single fiberoptic bronchoscopy during hospitalization according to clinical indications and with informed consent. During bronchoscopy, bronchoalveolar lavage (BAL) fluid samples will be collected for metagenomic, metabolomic, culture, biochemical, and cytological analyses. Additional mucosal biopsies will be obtained with separate consent if applicable.

Follow-up visits will include blood sample collection, sputum sampling (for cooperative children), spirometry, impulse oscillometry, and Fractional Exhaled Nitric Oxide measurements, without repeat bronchoscopy. The bronchoscopy procedure will not be repeated.

The study involves analysis of biological samples obtained during clinically indicated bronchoscopy, followed by a 5-year observation period. The findings will aid in distinguishing asthma phenotypes, identifying risk factors for asthma and protracted bacterial bronchitis, and improving the understanding of factors contributing to poor treatment response in these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age at the beginning of the study 0-17 years old
* Clinical indication and qualification by the attending physician for fiberoptic bronchoscopy under general anesthesia:

  * Obstruction of the airways:
  * Suspicion of foreign body aspiration
  * Persistent stridor
  * Abnormal result of functional tests of respiratory system - flattening of inspiratory or expiratory curve, presence of restriction (tested vital capacity <5 percentile) or irreversible obstruction (persistence of Tiffneau index <5 percentile despite administration of bronchodilators)
  * Radiological findings located in the course of the larynx, trachea or bronchi
  * Persistent atelectasis on subsequent radiological examinations
  * Persistent cough >4 weeks
  * Hemoptysis
  * Suspected laryngomalacia or tracheobronchomalacia
  * Suspected tracheoesophageal fistula
  * Persistent dyspnea unresponsive to anti-asthmatic treatment used for min. 2 months, with no other identifiable causes
  * Radiologically detected mediastinal abnormalities
  * Suspected presence of a vascular ring
  * Presence of excessive secretions that are impossible for the patient to expectorate
  * Fine needle biopsy of cystic lesions
* Obtained consent from patient/legal guardian for participation in the study

Exclusion Criteria:

* Active acute respiratory infection up to 4 weeks before the procedure
* Taking antibiotics or systemic glucocorticosteroids up to 4 weeks before the procedure
* Patients with very severe comorbidities (congenital immunodeficiencies, genetic disorders, neurological or neuromuscular diseases, cancer, severe congenital heart defects, heart failure, liver failure, inflammatory bowel disease, celiac disease)
* Patients with blood clotting disorders
* Children with diagnosed respiratory diseases other than asthma and protracted bacterial bronchitis - including interstitial diseases, tuberculosis, inflammation of small and medium-sized blood vessels
* Patients for whom >48 hours have passed between suspicion of foreign body aspiration and interventional bronchoscopy
* Children with foreign body aspiration having a foreign body located in the trachea

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited from among patients hospitalized in the University Clinical Center of the Medical University of Warsaw, Department of Pediatric Pulmonology and Allergology, and in the Medical University of Lodz, Department of Pediatric Pulmonology
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation on microbiome composition and diversity, cellular composition, and metabolomic profile between study groups | Index hospitalization, immediately after the procedure
  16S rRNA targeted sequencing, Shannon index, Chao1, and Pielou's evenness, Bray-Curtis dissimilarity, weighted UniFrac and unweighted UniFrac measures, PERMANOVA, principal coordinate analysis, ANCOM-BC2, ASVs tables generated by QIIME2 will be used as input for PICRUSt2 to infer functional profiles of the microbiomes, Biocrates' MetIDQ and MetaboAnalystR R package
Correlation of metagenomic and metabolomic findings on subsequent treatment and disease course between groups | 2 years
  16S rRNA targeted sequencing, Shannon index, Chao1, and Pielou's evenness, Bray-Curtis dissimilarity, weighted UniFrac and unweighted UniFrac measures, PERMANOVA, principal coordinate analysis, ANCOM-BC2, ASVs tables generated by QIIME2 will be used as input for PICRUSt2 to infer functional profiles of the microbiomes, Biocrates' MetIDQ and MetaboAnalystR R package, MANOVA and logistic regression, Cox proportional hazards model

SECONDARY OUTCOMES:
Comparison of the previous medical history and demographic characteristics across the study groups | At baseline
  MANOVA, neural networks and logistic regression
Assessment of the degree of asthma control among children diagnosed with asthma according to Global Initiative for Asthma | 5 years
  In children aged ≥5 years using the Asthma Control Questionnaire (ACQ) numeric scale, and in children <5 years using a questionnaire assessing the preceding month for asthma symptoms occurring more than twice per week, nocturnal cough or insomnia caused by dyspnea, need for short-acting β-mimetics more than twice per week, and physical activity limitations due to dyspnea.
Evaluation how the place of residence influences the incidence and clinical course of the studied diseases | 5 years
  Residence classified as urban (>100,000 inhabitants), town (<100,000 inhabitants), or rural area logistical regression
Assessment of exposure to PM10 dust at the place of residence during the year preceding study inclusion in children from each group | At baseline
  Data will be obtained from the Chief Environmental Protection Inspectorate website and will include average, minimum, and maximum monthly and annual concentrations, ANOVA/non-parametric tests
Comparison of the normalized difference vegetation index (NDVI) and chlorophyll index (CI) green levels between study groups at baseline | At baseline
  At place of residence
Comparison of the sputum culture at baseline and at the control visit | 2 years
  Comparison of fact of growth and number of CFU with Fisher's exact or χ² test
Comparison of the baseline sputum culture findings with BALF culture and metagenomic results | 2 years
  Comparison of fact of growth and number of CFU with Fisher's exact or χ² test, logistical regression
Evaluation of the initial Immunoglobulin E (IgE) concentrations and their dynamics of change between groups | 5 years
  Using medians with interquartile ranges and compared using the Mann-Whitney U or Kruskal-Wallis tests
Comparison of the eosinophil concentrations according to disease type and course | 5 years
  Using medians with interquartile ranges and compared using the Mann-Whitney U or Kruskal-Wallis tests
Assessment of the correlation between ICS used without an asthma diagnosis and airway dysbiosis | 2 years
  PERMANOVA and logistic regression
Evaluation of asthma treatment response, exacerbation rates, and need for bronchodilators according to airway metabolome profiles | 5 years
  PERMANOVA and logistic regression
Comparison of the asthma subtypes and evaluate possibilities for developing personalized treatment in selected pediatric groups | 2 years
  An attempt to assess the presence and relationship of asthma subtypes in relation to metagenomic and metabolomic findings PERMANOVA and logistic regression
Identification of the most common pathogens cultured from BALF samples in children with asthma, PBB, chronic cough, and in those taking ICS without an asthma diagnosis | Index hospitalization, immediately after the procedure
  descriptive statistics
Analysis of the frequency and type of antibiotic therapy in each study group and correlate these findings with the total number of respiratory diseases in individual participants. | 5 years
  Cox proportional hazards model
Evaluation of the recurrence rates of PBB and development of CSLD and BE based on identified airway pathogens | 5 years
  Cox proportional hazards model, descriptive statistics
Assessment of the prevalence of antibiotic-resistant strains among patients with PBB | 5 years
  descriptive statistics
Assessment of the time to PBB development in previously healthy children based on metagenomic and metabolomic findings | 5 years
  Cox proportional hazards model

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Feleszko, MD, PhD, Principal Investigator — Medical University of Warsaw

IPD SHARING:
Plan to Share IPD: No
IPD may be available upon request, by default IPD sharing is not planned.

REFERENCES:
- [Background] Martin J, Townshend J, Brodlie M. Diagnosis and management of asthma in children. BMJ Paediatr Open. 2022 Apr;6(1):e001277. doi: 10.1136/bmjpo-2021-001277. PMID 35648804
- [Background] Thomas R, Marchant JM, Goyal V, Masters IB, Yerkovich ST, Chang AB. Clinical utility of elective paediatric flexible bronchoscopy and impact on the quality of life: protocol for a single-centre, single-blind, randomised controlled trial. BMJ Open Respir Res. 2024 Feb 26;11(1):e001704. doi: 10.1136/bmjresp-2023-001704. PMID 38413121
- [Background] Licata MA, Mencarini P, Mastrobattista A, Carli SM, Cerva C, Mosti S, Libertone R, Zolezzi A, Vittozzi P, Nisii C, Mazzarelli A, Cannas A, Navarra A, Ianniello S, Trisolini R, Goletti D, Palmieri F, Gualano G. Clinical Utility of Induced Sputum and Bronchoalveolar Lavage Cultures in Diagnosing Nontuberculous Mycobacterial Pulmonary Disease. Pathogens. 2024 Dec 3;13(12):1064. doi: 10.3390/pathogens13121064. PMID 39770324
- [Background] Chang AB, Upham JW, Masters IB, Redding GR, Gibson PG, Marchant JM, Grimwood K. Protracted bacterial bronchitis: The last decade and the road ahead. Pediatr Pulmonol. 2016 Mar;51(3):225-42. doi: 10.1002/ppul.23351. Epub 2015 Dec 4. PMID 26636654
- [Background] Gallucci M, Pedretti M, Giannetti A, di Palmo E, Bertelli L, Pession A, Ricci G. When the Cough Does Not Improve: A Review on Protracted Bacterial Bronchitis in Children. Front Pediatr. 2020 Aug 7;8:433. doi: 10.3389/fped.2020.00433. eCollection 2020. PMID 32850546
- [Background] Weiss AJ, Liang L, Martin K. Overview of Hospital Stays Among Children and Adolescents, 2019. 2022 Nov 29. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #299. Available from http://www.ncbi.nlm.nih.gov/books/NBK588376/ PMID 36622925
- [Background] Levy ML, Fleming L, Warner JO, Bush A. Paediatric asthma care in the UK: fragmented and fatally fallible. Br J Gen Pract. 2019 Aug;69(685):405-406. doi: 10.3399/bjgp19X704933. No abstract available. PMID 31345822
- [Background] Januska MN, Goldman DL, Webley W, Teague WG, Cohen RT, Bunyavanich S, Vicencio AG. Bronchoscopy in severe childhood asthma: Irresponsible or irreplaceable? Pediatr Pulmonol. 2020 Mar;55(3):795-802. doi: 10.1002/ppul.24569. Epub 2019 Nov 15. PMID 31730298
- [Background] Zhang J, Wurzel DF, Perret JL, Lodge CJ, Walters EH, Dharmage SC. Chronic Bronchitis in Children and Adults: Definitions, Pathophysiology, Prevalence, Risk Factors, and Consequences. J Clin Med. 2024 Apr 20;13(8):2413. doi: 10.3390/jcm13082413. PMID 38673686
- [Background] Escribano Montaner A, Garcia de Lomas J, Villa Asensi JR, Asensio de la Cruz O, de la Serna Blazquez O, Santiago Burruchaga M, Mondejar Lopez P, Torrent Vernetta A, Feng Y, Van Dyke MK, Reyes J, Garcia-Corbeira P, Talarico CA; EPI-Strep-064 study group. Bacteria from bronchoalveolar lavage fluid from children with suspected chronic lower respiratory tract infection: results from a multi-center, cross-sectional study in Spain. Eur J Pediatr. 2018 Feb;177(2):181-192. doi: 10.1007/s00431-017-3044-3. Epub 2017 Dec 29. PMID 29285648
- [Background] Chang AB, Bell SC, Byrnes CA, Dawkins P, Holland AE, Kennedy E, King PT, Laird P, Mooney S, Morgan L, Parsons M, Poot B, Toombs M, Torzillo PJ, Grimwood K. Thoracic Society of Australia and New Zealand (TSANZ) position statement on chronic suppurative lung disease and bronchiectasis in children, adolescents and adults in Australia and New Zealand. Respirology. 2023 Apr;28(4):339-349. doi: 10.1111/resp.14479. Epub 2023 Mar 2. PMID 36863703
- [Background] Wiltingh H, Marchant JM, Goyal V. Cough in Protracted Bacterial Bronchitis and Bronchiectasis. J Clin Med. 2024 Jun 4;13(11):3305. doi: 10.3390/jcm13113305. PMID 38893016
- [Background] Marsh RL, Smith-Vaughan HC, Chen ACH, Marchant JM, Yerkovich ST, Gibson PG, Pizzutto SJ, Hodge S, Upham JW, Chang AB. Multiple Respiratory Microbiota Profiles Are Associated With Lower Airway Inflammation in Children With Protracted Bacterial Bronchitis. Chest. 2019 Apr;155(4):778-786. doi: 10.1016/j.chest.2019.01.002. Epub 2019 Jan 17. PMID 30660785
- [Background] Broderick DTJ, Waite DW, Marsh RL, Camargo CA Jr, Cardenas P, Chang AB, Cookson WOC, Cuthbertson L, Dai W, Everard ML, Gervaix A, Harris JK, Hasegawa K, Hoffman LR, Hong SJ, Josset L, Kelly MS, Kim BS, Kong Y, Li SC, Mansbach JM, Mejias A, O'Toole GA, Paalanen L, Perez-Losada M, Pettigrew MM, Pichon M, Ramilo O, Ruokolainen L, Sakwinska O, Seed PC, van der Gast CJ, Wagner BD, Yi H, Zemanick ET, Zheng Y, Pillarisetti N, Taylor MW. Bacterial Signatures of Paediatric Respiratory Disease: An Individual Participant Data Meta-Analysis. Front Microbiol. 2021 Dec 23;12:711134. doi: 10.3389/fmicb.2021.711134. eCollection 2021. PMID 35002989
- [Background] Ausejo M, Saenz A, Pham B, Kellner JD, Johnson DW, Moher D, Klassen TP. The effectiveness of glucocorticoids in treating croup: meta-analysis. BMJ. 1999 Sep 4;319(7210):595-600. doi: 10.1136/bmj.319.7210.595. PMID 10473471
- [Background] Oymar K, Mikalsen IB, Furu K, Nystad W, Karlstad O. Prescription patterns of inhaled corticosteroids for preschool children--A Norwegian register study. Pediatr Allergy Immunol. 2015 Nov;26(7):655-61. doi: 10.1111/pai.12429. Epub 2015 Jul 14. PMID 26110251
- [Background] Hartmann JE, Albrich WC, Dmitrijeva M, Kahlert CR. The Effects of Corticosteroids on the Respiratory Microbiome: A Systematic Review. Front Med (Lausanne). 2021 Mar 10;8:588584. doi: 10.3389/fmed.2021.588584. eCollection 2021. PMID 33777968
- [Background] Contoli M, Pauletti A, Rossi MR, Spanevello A, Casolari P, Marcellini A, Forini G, Gnesini G, Marku B, Barnes N, Rizzi A, Curradi G, Caramori G, Morelli P, Papi A. Long-term effects of inhaled corticosteroids on sputum bacterial and viral loads in COPD. Eur Respir J. 2017 Oct 5;50(4):1700451. doi: 10.1183/13993003.00451-2017. Print 2017 Oct. PMID 28982774
- [Background] Bergmann M, Haasenritter J, Beidatsch D, Schwarm S, Horner K, Bosner S, Grevenrath P, Schmidt L, Viniol A, Donner-Banzhoff N, Becker A. Prevalence, aetiologies and prognosis of the symptom cough in primary care: a systematic review and meta-analysis. BMC Fam Pract. 2021 Jul 12;22(1):151. doi: 10.1186/s12875-021-01501-0. PMID 34253179
- [Background] Chang AB, Oppenheimer JJ, Irwin RS; CHEST Expert Cough Panel. Managing Chronic Cough as a Symptom in Children and Management Algorithms: CHEST Guideline and Expert Panel Report. Chest. 2020 Jul;158(1):303-329. doi: 10.1016/j.chest.2020.01.042. Epub 2020 Mar 14. PMID 32179109
- [Background] Chantzaras AP, Panagiotou P, Karageorgos S, Douros K. A systematic review of using flexible bronchoscopy to remove foreign bodies from paediatric patients. Acta Paediatr. 2022 Jul;111(7):1301-1312. doi: 10.1111/apa.16351. Epub 2022 Apr 12. PMID 35388522
- [Background] Cramer N, Jabbour N, Tavarez MM, Taylor RS. Foreign Body Aspiration(Archived). 2023 Jul 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK531480/ PMID 30285375
- [Background] Davidson KR, Ha DM, Schwarz MI, Chan ED. Bronchoalveolar lavage as a diagnostic procedure: a review of known cellular and molecular findings in various lung diseases. J Thorac Dis. 2020 Sep;12(9):4991-5019. doi: 10.21037/jtd-20-651. PMID 33145073
- [Background] Hachim MY, Elemam NM, Ramakrishnan RK, Salameh L, Olivenstein R, Hachim IY, Venkatachalam T, Mahboub B, Al Heialy S, Halwani R, Hamid Q, Hamoudi R. Blood and Salivary Amphiregulin Levels as Biomarkers for Asthma. Front Med (Lausanne). 2020 Oct 29;7:561866. doi: 10.3389/fmed.2020.561866. eCollection 2020. PMID 33195308
- [Background] Doeing DC, Solway J. Airway smooth muscle in the pathophysiology and treatment of asthma. J Appl Physiol (1985). 2013 Apr;114(7):834-43. doi: 10.1152/japplphysiol.00950.2012. Epub 2013 Jan 10. PMID 23305987
- [Background] Muller L, Brighton LE, Carson JL, Fischer WA 2nd, Jaspers I. Culturing of human nasal epithelial cells at the air liquid interface. J Vis Exp. 2013 Oct 8;(80):50646. doi: 10.3791/50646. PMID 24145828
- [Background] Bolyen E, Rideout JR, Dillon MR, Bokulich NA, Abnet CC, Al-Ghalith GA, Alexander H, Alm EJ, Arumugam M, Asnicar F, Bai Y, Bisanz JE, Bittinger K, Brejnrod A, Brislawn CJ, Brown CT, Callahan BJ, Caraballo-Rodriguez AM, Chase J, Cope EK, Da Silva R, Diener C, Dorrestein PC, Douglas GM, Durall DM, Duvallet C, Edwardson CF, Ernst M, Estaki M, Fouquier J, Gauglitz JM, Gibbons SM, Gibson DL, Gonzalez A, Gorlick K, Guo J, Hillmann B, Holmes S, Holste H, Huttenhower C, Huttley GA, Janssen S, Jarmusch AK, Jiang L, Kaehler BD, Kang KB, Keefe CR, Keim P, Kelley ST, Knights D, Koester I, Kosciolek T, Kreps J, Langille MGI, Lee J, Ley R, Liu YX, Loftfield E, Lozupone C, Maher M, Marotz C, Martin BD, McDonald D, McIver LJ, Melnik AV, Metcalf JL, Morgan SC, Morton JT, Naimey AT, Navas-Molina JA, Nothias LF, Orchanian SB, Pearson T, Peoples SL, Petras D, Preuss ML, Pruesse E, Rasmussen LB, Rivers A, Robeson MS 2nd, Rosenthal P, Segata N, Shaffer M, Shiffer A, Sinha R, Song SJ, Spear JR, Swafford AD, Thompson LR, Torres PJ, Trinh P, Tripathi A, Turnbaugh PJ, Ul-Hasan S, van der Hooft JJJ, Vargas F, Vazquez-Baeza Y, Vogtmann E, von Hippel M, Walters W, Wan Y, Wang M, Warren J, Weber KC, Williamson CHD, Willis AD, Xu ZZ, Zaneveld JR, Zhang Y, Zhu Q, Knight R, Caporaso JG. Reproducible, interactive, scalable and extensible microbiome data science using QIIME 2. Nat Biotechnol. 2019 Aug;37(8):852-857. doi: 10.1038/s41587-019-0209-9. No abstract available. PMID 31341288
- [Background] Lin H, Peddada SD. Multigroup analysis of compositions of microbiomes with covariate adjustments and repeated measures. Nat Methods. 2024 Jan;21(1):83-91. doi: 10.1038/s41592-023-02092-7. Epub 2023 Dec 29. PMID 38158428
- [Background] Douglas GM, Maffei VJ, Zaneveld JR, Yurgel SN, Brown JR, Taylor CM, Huttenhower C, Langille MGI. PICRUSt2 for prediction of metagenome functions. Nat Biotechnol. 2020 Jun;38(6):685-688. doi: 10.1038/s41587-020-0548-6. No abstract available. PMID 32483366
- [Background] Pang Z, Xu L, Viau C, Lu Y, Salavati R, Basu N, Xia J. MetaboAnalystR 4.0: a unified LC-MS workflow for global metabolomics. Nat Commun. 2024 May 1;15(1):3675. doi: 10.1038/s41467-024-48009-6. PMID 38693118